CLINICAL TRIAL: NCT05108909
Title: Rapid Diagnosis and Prognosis Recognition of Imaging and Biomarkers in Mild to Moderate Traumatic Brain Injury
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: First Affiliated Hospital Xi'an Jiaotong University (Other)
Collaborators: Xi'an Jiaotong University (Other); Second Affiliated Hospital of Wenzhou Medical University (Other); Central South University (Other); Xijing Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 82071993-2
Record Dates: First submitted 2021-09-24; First posted 2021-11-05 (Actual); Last update posted 2022-01-04 (Actual); Status verified 2021-10

CONDITIONS: MTBI - Mild Traumatic Brain Injury; Moderate Traumatic Brain Injury
Keywords: mild to moderate traumatic brain injury; biomarkers; magnetic resonance image; CT; diagnosis; Prognostic identification
MeSH Terms: conditions — Brain Concussion; Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — whole blood, gut microbiota, urine
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- mild to moderate traumatic brain injury: patients diagnosed with mild to moderate traumatic brain injury within 1 week after onset of TBI.
  Interventions: Device: MRI, CT, and serum biomarkers
- isolated orthopaedic trauma patients: Patients with isolated orthopaedic trauma were identified and enrolled using the same process as that for patients with TBI.
  Interventions: Device: MRI, CT, and serum biomarkers
- healthy non-injury control: Healthy non-injured controls were recruited either via a relationship with a TRACK-TBI participant or through public advertisement within TRACK-TBI institutions, and were able to provide informed consent.
  Interventions: Device: MRI, CT, and serum biomarkers

INTERVENTIONS:
Device: MRI, CT, and serum biomarkers — magnetic resonance image Imaging data were collected in a strong magnetic field, and collected the serum of participants.

SUMMARY:
The investigators will carry out multi-center and large sample research based on the Chinese population, screen the optimal diagnostic and prognosis recognition biomarkers and analyze the diagnostic critical cutoff values in patients with mild to moderate traumatic brain injury, so as to provide a substantial basis for clinical diagnosis and prognosis recognition.

DETAILED DESCRIPTION:
Traumatic brain injury (TBI) is a complex disorder that comprises a spectrum of intracranial pathologies, many of which present diagnostic challenges. Detection of intracranial injuries after TBI relies on head CT, which is overused and resource intensive. Prior studies have shown the potential for blood-based brain injury biomarkers to predict the absence of intracranial injury after TBI and aid in reducing unnecessary head CT use. Furthermore, plasma biomarker concentrations in the acute phase after TBI identified patients with a suspected TBI and normal head CT who had detectable pathology on MRI. However, most of the current studies are based on the European and American population, and whether the research results are applicable to the Chinese population remains to be studied. Therefore, the investigators will carry out multi-center and large sample research based on the Chinese population, screen the optimal diagnostic and prognosis recognition biomarkers and analyze the diagnostic critical cutoff values, so as to provide a substantial basis for clinical diagnosis and prognosis recognition.

ELIGIBILITY:
Inclusion Criteria:

* age 18-75 years at time of recruitment.
* Glasgow Coma Scale (GCS) score of 9-15 at the time of informed consent.
* non-penetrating TBI resulting from an external force.
* diagnosed within 1 week after onset of TBI.
* provision of informed written consent.

Exclusion Criteria:

* acute suspected stroke, neurosurgery, stroke or TIA within the last 30 days.
* neurodegenerative disease or other neurological disorder including dementia, Parkinson's disease, multiple sclerosis, seizure disorder, brain tumors.
* a history of a previous brain injury, or a history of concurrent substance or alcohol abuse;
* the manifestation of TBI caused by medications, alcohol, drugs for other injuries (such as systemic injuries, facial injuries, or intubation).
* pregnancy or breastfeeding.
* Patients with contraindications to MRI scanning (such as patients with metal implants in their bodies, cardiac pacemakers, dentures, etc.)
* participation in a clinical research study with potential to affect the results of this study

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: TBI patients will be recruited from the emergency department of hospital.
Sampling Method: Probability Sample
Enrollment: 800 (Estimated)
Dates: Start 2021-09-01 (Actual); Primary Completion 2025-08-31 (Estimated); Study Completion 2025-08-31 (Estimated)

PRIMARY OUTCOMES:
The concentration of serum biomarkers. | baseline (early injury), post-traumatic for 3 months, 6 months, and 12 months.
  the concentration of GFAP with pg/mL, S-100B with pg/mL，IL-6 with pg/mL, IL-8 with pg/mL, IL-10 with pg/mL, IL-1β with pg/mL, TNF-α with pg/mL, UCH-L1 with pg/mL, NSE with pg/mL, T-Tau with pg/mL, P-Tau with pg/mL, NFL with pg/mL, BDNF with pg/mL, and VEGF with pg/mL;
Score of Extended Glasgow Outcome Scale. | post-traumatic for 3 months
  The functional outcome of TBI patients. The minimum value is 1, and the maximum value is 8. The higher scores mean a better outcome.
Score of Extended Glasgow Outcome Scale. | post-traumatic for 6 months
  The functional outcome of TBI patients. The minimum value is 1, and the maximum value is 8. The higher scores mean a better outcome.
Score of Extended Glasgow Outcome Scale. | post-traumatic for 12 months
  The functional outcome of TBI patients. The minimum value is 1, and the maximum value is 8. The higher scores mean a better outcome.
Number of participants with positive head CT scan | baseline (early injury)
  CT-positive was defined as the presence of one or more of the following injuries: acute epidural haematoma, acute subdural haematoma, indeterminate extraaxial haemorrhage, intraventricular haemorrhage, parenchymal haematoma, petechial haemorrhagic or bland sheer injury, subarachnoid haemorrhage, brain oedema, brain herniation, non-haemorrhagic contusion, ventricular compression, ventricular trapping, cranial fractures, depressed skull fractures, facial fractures, scalp injury, or skull base fractures.
Number of participants with MRI abnormalities | baseline (early injury)
  MRI abnormalities were quantified according to common data elements standards and definitions by three board-certified neuroradiologists masked to the identity and clinical history of the patient. MRI scans were read as positive if there was evidence of acute intracranial pathology consistent with TBI (eg, contusion, traumatic axonal injury, diffuse axonal injury).

SECONDARY OUTCOMES:
Change from baseline brain structure measures at 3 months | baseline (early injury), post-traumatic for 3 months.
  The changes of brain volume (mm3) are evaluated by structural MRI
Change from baseline brain structure measures at 6 months | baseline (early injury), post-traumatic for 6 months.
  The changes of brain volume (mm3) are evaluated by structural MRI
Change from baseline brain structure measures at 12 months | baseline (early injury), post-traumatic for 12 months.
  The changes of brain volume (mm3) are evaluated by structural MRI
White matter integrity at baseline (early injury), post-traumatic for 3 months,6 months, and 12 months. | baseline (early injury), post-traumatic for 3 months,6 months, and 12 months.
  The white matter integrity are characterized by fractional anisotropy (FA) which calculated by diffusion tensor imaging.

CONTACTS AND LOCATIONS:
Overall Officials: Ming Zhang, phD, Principal Investigator — First Affiliated Hospital of Xian Jiaotong University
Locations (1):
- First Affiliated Hospital of Xian Jiaotong University, Xi'an, Shaanxi, China